CLINICAL TRIAL: NCT00880763
Title: A Phase II Randomized Placebo-controlled Study to Evaluate the Safety and Efficacy of MK-7009 Administered Concomitantly With Pegylated-Interferon and Ribavirin for 28 Days in Japanese Treatment-Experienced Patients With Chronic Hepatitis C Infection
Brief Title: A Study of Safety and Efficacy of Vaniprevir Administered With Pegylated-Interferon and Ribavirin in Japanese Participants With Chronic Hepatitis C Infection (7009-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7009-016; 2009_576
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — vaniprevir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vaniprevir 200 mg + peg-IFN + ribavirin (Experimental): Participants will receive vaniprevir 100 mg twice daily in combination with peg-IFN and ribavirin for 28 days. Participants will continue peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
  Interventions: Drug: Vaniprevir; Drug: Pegylated Interferon (peg-IFN); Drug: Ribavirin
- Vaniprevir 600 mg + peg-IFN + ribavirin (Experimental): Participants will receive vaniprevir 300 mg twice daily in combination with peg-IFN and ribavirin for 28 days. Participants will continue peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
  Interventions: Drug: Vaniprevir; Drug: Pegylated Interferon (peg-IFN); Drug: Ribavirin
- Vaniprevir 1200 mg + peg-IFN + ribavirin (Experimental): Participants will receive vaniprevir 600 mg twice daily in combination with peg-IFN and ribavirin for 28 days. Participants will continue peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
  Interventions: Drug: Vaniprevir; Drug: Pegylated Interferon (peg-IFN); Drug: Ribavirin
- Placebo + peg-IFN + ribavirin (Placebo Comparator): Participants will receive placebo twice daily in combination with peg-IFN and ribavirin for 28 days. Participants will continue peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
  Interventions: Drug: Pegylated Interferon (peg-IFN); Drug: Ribavirin; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Vaniprevir — Vaniprevir oral capsule administered twice daily (200, 600 or 1200 mg/day) for 28 days
  Other Names: MK7009
  Arms: Vaniprevir 1200 mg + peg-IFN + ribavirin; Vaniprevir 200 mg + peg-IFN + ribavirin; Vaniprevir 600 mg + peg-IFN + ribavirin
Drug: Pegylated Interferon (peg-IFN) — Open-label peg-IFN alfa-2a subcutaneous injection (sourced locally) administered weekly, 180 micrograms, for 6 weeks
Drug: Ribavirin — Open-label ribavirin (sourced locally) administered orally twice daily, 600 to 1000 mg/day, for 6 weeks
Drug: Comparator: Placebo — Placebo to vaniprevir oral capsule twice daily for 28 days
  Arms: Placebo + peg-IFN + ribavirin

SUMMARY:
The study evaluates safety and efficacy of vaniprevir (MK7009), when administered with Pegylated-Interferon (peg-IFN) and Ribavirin, in Japanese patients with Hepatitis C infection. The primary hypotheses are that 1.) the proportion of patients achieving rapid viral response (RVR) in one or more of the vaniprevir treatment groups is superior to that in the placebo group, when each is administered concomitantly with pegylated interferon (peg-IFN) α-2a and ribavirin; and 2.) vaniprevir at the studied doses is well tolerated compared with placebo, when each is administered concomitantly with peg-IFN α-2a and ribavirin for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Has chronic genotype 1 Hepatitis C infection

Exclusion Criteria:

* Has not tolerated previous course of peg-IFN and ribavirin
* Has HIV
* Has Hepatitis B
* Has a history of clinically significant medical condition that may interfere with the study (e.g., stroke or chronic seizures or major neurological disorder) or is contraindicated for treatment with peg-IFN and ribavirin

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-04-20 (Actual); Primary Completion 2010-06-03 (Actual); Study Completion 2012-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hayashi N, Mobashery N, Izumi N. Vaniprevir plus peginterferon alfa-2a and ribavirin in treatment-experienced Japanese patients with hepatitis C virus genotype 1 infection: a randomized phase II study. J Gastroenterol. 2015 Feb;50(2):238-48. doi: 10.1007/s00535-014-0979-2. Epub 2014 Aug 13. PMID 25115901
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-016&kw=7009-016&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initial treatment period (Part 1) includes up through Week 6; Extension period (Part 2) includes from Week 6 through Week 96.
Groups:
- Vaniprevir 200 mg + Peg-IFN + Ribavirin: Participants received vaniprevir 100 mg twice daily in combination with peg-IFN and ribavirin for 28 days. Participants continued peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
- Vaniprevir 600 mg + Peg-IFN + Ribavirin: Participants received vaniprevir 300 mg twice daily in combination with peg-IFN and ribavirin for 28 days. Participants continued peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
- Vaniprevir 1200 mg + Peg-IFN + Ribavirin: Participants received vaniprevir 600 mg twice daily in combination with peg-IFN and ribavirin for 28 days. Participants continued peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
- Placebo + Peg-IFN + Ribavirin: Participants received placebo twice daily in combination with peg-IFN and ribavirin for 28 days. Participants continued peg-IFN and ribavirin through Week 6 or, at the investigators discretion, up to Week 72.
Period: Initial Treatment Period (Part 1)
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Started | 23 | 22 | 23 | 22
Completed | 23 | 22 | 23 | 22
Not Completed | 0 | 0 | 0 | 0
Period: Extension Period (Part 2)
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Started | 23 | 22 | 23 | 22
Completed | 23 | 19 | 20 | 19
Not Completed | 0 | 3 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin | Total
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (6.5) | 54.3 (7.6) | 56.3 (7.8) | 54.7 (6.9) | 55.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 12 | 14 | 45
  Male | 11 | 15 | 11 | 8 | 45
Region of Enrollment [Number; unit: Participants]
  Japan | 23 | 22 | 23 | 22 | 90
Genotype [Number; unit: Participants]
  Genotype 1a | 1 | 1 | 0 | 1 | 3
  Genotype 1b | 22 | 21 | 23 | 21 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Rapid Viral Response
Description: Rapid viral response (RVR) is defined as undetectable hepatitis C virus ribonucleic acid (HCV RNA) at Week 4. Serum HCV RNA levels were measured using Roche COBAS TaqMan HCV Auto assay. The limit of quantification was 1.2 log IU/mL (15 IU/mL) and the limit of detection was <1.2 log IU/mL, but with no specific value. The Data-As-Observed (DAO) approach was used to handle missing data.
Time Frame: Week 4
Population: Per protocol population excludes participants for important deviations from the protocol that may substantially affect the results of the primary efficacy analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Number analyzed (Participants) | 22 | 20 | 21 | 20
Percentage of participants | 86.4 | 95.0 | 76.2 | 20.0
Statistical Analysis 1: Comparison: Vaniprevir 200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Adjusted difference in percent = 65.1, 95% CI 2-sided [37.0 to 82.8] — Computed using Miettinen and Nurminen method adjusting the strata (participation of Intensive-pharmacokinetic cohort vs. not)
Statistical Analysis 2: Comparison: Vaniprevir 600 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Adjusted difference in percent = 74.5, 95% CI 2-sided [47.6 to 89.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Vaniprevir 1200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Adjusted difference in percent = 55.4, 95% CI 2-sided [24.9 to 76.0] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Achieving a > or = 2-log10 Decrease in HCV RNA From Baseline to Week 4
Description: Serum HCV RNA levels were measured using Roche COBAS TaqMan HCV Auto assay. The DAO approach was used to handle missing data.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Number analyzed (Participants) | 22 | 20 | 21 | 20
Percentage of participants | 100 | 100 | 100 | 95
Statistical Analysis 1: Comparison: Vaniprevir 200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Adjusted difference in percent = 4.8, 95% CI 2-sided [-11.3 to 24.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vaniprevir 600 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Adjusted difference in percent = 4.9, 95% CI 2-sided [-12.4 to 24.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Vaniprevir 1200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Adjusted difference in percent = 4.8, 95% CI 2-sided [-12.0 to 24.2] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Achieving a > or = 3-log10 Decrease in HCV RNA From Baseline to Week 4
Description: as for outcome 2
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Number analyzed (Participants) | 22 | 20 | 21 | 20
Percentage of participants | 100 | 100 | 100 | 85
Statistical Analysis 1: Comparison: Vaniprevir 200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Adjusted difference in percent = 14.5, 95% CI 2-sided [-2.5 to 36.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vaniprevir 600 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Adjusted difference in percent = 14.6, 95% CI 2-sided [-3.4 to 36.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Vaniprevir 1200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Adjusted difference in percent = 14.4, 95% CI 2-sided [-3.3 to 36.1] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in HCV RNA in log10 at Week 4
Description: Change from baseline in HCV RNA at Week 4 was calculated by subtracting Week 4 HCV RNA level from Baseline HCV RNA level. HCV RNA is measured as International Units per milliliter (IU/mL). Serum HCV RNA levels were measured using Roche COBAS TaqMan HCV Auto assay. The DAO approach was used to handle missing data.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL in Log10
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Number analyzed (Participants) | 22 | 20 | 21 | 20
IU/mL in Log10
  Baseline | 6.6 (0.6) [-6.8 to -6.1] | 6.6 (0.6) [-7.0 to -6.2] | 6.6 (0.8) [-6.7 to -6.0] | 6.6 (0.5) [-5.1 to -4.3]
  Change from Baseline | -6.5 (0.6) | -6.6 (0.6) | -6.3 (0.8) | -4.7 (1.6)
Statistical Analysis 1: Comparison: Vaniprevir 200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Difference in least squares mean = -1.8, 95% CI 2-sided [-2.3 to -1.2] — Computed using a longitudinal data analysis model including treatment, time and the interaction of time by treatment, with a restriction of the same baseline mean across treatment groups
Statistical Analysis 2: Comparison: Vaniprevir 600 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Difference in least squares mean = -1.9, 95% CI 2-sided [-2.4 to -1.3] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Vaniprevir 1200 mg + Peg-IFN + Ribavirin vs Placebo + Peg-IFN + Ribavirin; Test type: Superiority or Other; Difference in least squares mean = -1.6, 95% CI 2-sided [-2.2 to -1.1] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: Up to 6 weeks
Population: The All Participants as Treated population consists of all randomized participants who received at least one dose of study treatment. Participants are included in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: Participants
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Number analyzed (Participants) | 23 | 22 | 23 | 22
Participants | 23 | 22 | 23 | 22

6. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 5
Time Frame: Up to 6 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Number analyzed (Participants) | 23 | 22 | 23 | 22
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: up to 6 weeks (Part 1 only); Serious adverse events: up to 96 weeks (Parts 1 and 2 including 24-week follow-up period)
Description: All participants as treated population consists of all randomized participants who received at least one dose of study. Participants are included in the treatment group corresponding to the study treatment they actually received.
Arm/Group | Vaniprevir 200 mg + Peg-IFN + Ribavirin | Vaniprevir 600 mg + Peg-IFN + Ribavirin | Vaniprevir 1200 mg + Peg-IFN + Ribavirin | Placebo + Peg-IFN + Ribavirin
Serious Adverse Events (participants affected / at risk) | 2/23 | 2/22 | 0/23 | 2/22
Other Adverse Events (participants affected / at risk) | 23/23 | 22/22 | 23/23 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 200 mg + Peg-IFN + Ribavirin (N=23) | Vaniprevir 600 mg + Peg-IFN + Ribavirin (N=22) | Vaniprevir 1200 mg + Peg-IFN + Ribavirin (N=23) | Placebo + Peg-IFN + Ribavirin (N=22)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaniprevir 200 mg + Peg-IFN + Ribavirin (N=23) | Vaniprevir 600 mg + Peg-IFN + Ribavirin (N=22) | Vaniprevir 1200 mg + Peg-IFN + Ribavirin (N=23) | Placebo + Peg-IFN + Ribavirin (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 3 (3) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 6 (6) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 5 (5) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 6 (7) | 3 (3) | 3 (4)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 9 (9) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 9 (9) | 4 (4)
Periodontitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Fatigue (General disorders) | 7 (7) | 2 (2) | 6 (6) | 4 (5)
Feeling hot (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Malaise (General disorders) | 2 (2) | 3 (3) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 12 (13) | 15 (15) | 9 (10) | 12 (15)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Eosinophil count decreased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 6 (6)
Haematocrit decreased (Investigations) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Haemoglobin decreased (Investigations) | 9 (9) | 7 (7) | 10 (10) | 8 (8)
Monocyte count increased (Investigations) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (7) | 9 (9) | 11 (13) | 7 (7)
Platelet count decreased (Investigations) | 12 (12) | 11 (13) | 9 (10) | 9 (9)
White blood cell count decreased (Investigations) | 15 (15) | 15 (15) | 15 (15) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 8 (12) | 2 (2) | 9 (10) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 3 (3) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.